CLINICAL TRIAL: NCT03829501
Title: A Phase 1/2, Open-label, Multi-center Study of the Safety and Efficacy of KY1044 as Single Agent and in Combination With Anti-PD-L1 (Atezolizumab) in Adult Patients With Selected Advanced Malignancies
Brief Title: A Phase 1/2, Open-label, Multi-center Study of the Safety and Efficacy of Alomfilimab (KY1044) as Single Agent and in Combination With Anti-PD-L1 (Atezolizumab) in Adult Patients With Selected Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early discontinuation based on strategic sponsor decision not driven by any safety concerns.
Sponsor: Kymab Limited (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY1044-CT01; Sanofi Study ID (Other: TCD17370); 2018-003172-12 (EudraCT Number); U1111-1269-6777 (Other: WHO ICTRP)
Record Dates: First submitted 2019-01-17; First posted 2019-02-04 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Non-small Cell Lung Cancer; Hepatocellular Carcinoma; Esophageal Cancer; Gastric Cancer; Melanoma; Renal Cell Carcinoma; Pancreatic Cancer; Cervical Cancer; Triple Negative Breast Cancer; Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Carcinoma, Hepatocellular; Esophageal Neoplasms; Stomach Neoplasms; Melanoma; Carcinoma, Renal Cell; Pancreatic Neoplasms; Uterine Cervical Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Alomfilimab Monotherapy (Experimental): Participants will receive alomfilimab 0.8 to 240 mg as a single agent via intravenous (IV) infusion every 3 weeks (Q3W).
  Interventions: Drug: Alomfilimab
- Phase 1: Alomfilimab + Atezolizumab Combination Therapy (Experimental): Participants will receive alomfilimab 2.4 to 80 mg in combination with atezolizumab 1200 mg via IV infusion Q3W.
  Interventions: Drug: Alomfilimab; Drug: Atezolizumab
- Phase 2: Alomfilimab + Atezolizumab in Anti-PD-(L)1 Naïve Participants (Experimental): Anti-PD-(L)1 naïve participants with pancreatic cancer, triple negative breast cancer (BC) or head and neck squamous cell carcinoma (HNSCC) will receive alomfilimab 2.4 to 24 mg in combination with atezolizumab 1200 mg via IV infusion Q3W.
  Interventions: Drug: Alomfilimab; Drug: Atezolizumab
- Phase 2: Alomfilimab + Atezolizumab in Pre-treated Participants (Experimental): Pre-treated participants with pancreatic cancer, triple negative BC or HNSCC will receive alomfilimab 2.4 to 24 mg in combination with atezolizumab 1200 mg via IV infusion Q3W.
  Interventions: Drug: Alomfilimab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Alomfilimab — A human anti-ICOS monoclonal antibody
  Other Names: KY1044; SAR445256
Drug: Atezolizumab — An anti-PD-L1 monoclonal antibody
  Other Names: TECENTRIQ
  Arms: Phase 1: Alomfilimab + Atezolizumab Combination Therapy; Phase 2: Alomfilimab + Atezolizumab in Anti-PD-(L)1 Naïve Participants; Phase 2: Alomfilimab + Atezolizumab in Pre-treated Participants

SUMMARY:
A Phase 1/2, open label, multi-center study to evaluate the safety, efficacy and tolerability of alomfilimab as single agent and in combination with anti-PD-L1 (atezolizumab) in adult patients with selected advanced malignancies, who are ineligible for or there are no available therapies known to confer a clinical benefit for their disease, or they have exhausted all such available options in each indication and therefore will be patients for whom a clinical trial is appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years (≥20 years in Taiwan)
* Histologically documented advanced/metastatic malignancies
* Phase 1 and Phase 2 participants with advanced/metastatic malignancies who have measurable disease (non-measurable disease is allowed only in Phase 1) as determined by RECIST 1.1 will be eligible if, according to the National Comprehensive Cancer Network (NCCN) guidelines, there are no available therapies known to confer a clinical benefit for their disease, or they have exhausted all such available options. Additionally, the following specific tumor indications will be enrolled:

  1. Phase 1: Participants with advanced/metastatic malignancies, and preferred indications (non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), hepatocellular carcinoma (HCC), melanoma, cervical, esophageal, gastric, renal, pancreatic, and triple negative breast cancer)
  2. Phase 2 Alomfilimab single agent: Participants with advanced/metastatic malignancies in indications in which signs of anti-tumor activity (Complete Response (CR), Partial Response (PR) or durable stable disease (SD) with tumor shrinkage that does not qualify for PR) were seen during the dose escalation of Alomfilimab as single agent
  3. Phase 2 Alomfilimab in combination with atezolizumab: Participants with advanced/metastatic malignancies in the selected indications below, and/or indications which have shown promising activity in Phase 1:

     * NSCLC (anti-PD-(L)1 therapy naïve and pre-treated between 1 and 2 prior lines of systemic therapy for advanced disease)
     * Gastric (anti-PD-(L)1 therapy naïve and pre-treated)
     * Recurrent and/or metastatic HNSCC (anti-PD-(L)1 therapy naïve and pre-treated between 1 and 2 prior lines of systemic therapy for advanced disease)
     * Esophageal (anti-PD-(L)1 therapy naïve and pre-treated)
     * Cervical (anti-PD-(L)1 therapy naïve and pre-treated)
     * Indications, in which signs of anti-tumor activity has been observed in Phase 1 with Alomfilimab in combination with atezolizumab
* Prior therapy with anti-PD-(L)1 inhibitors is allowed provided any toxicity attributed to prior anti-PD-(L)1-directed therapy did not lead to discontinuation of therapy
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Life expectancy longer than 12 weeks
* Must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Participants must be willing to undergo a new tumor biopsy at screening, and during therapy on the study

Exclusion Criteria:

* Presence of symptomatic central nervous system (CNS) metastases, or CNS metastases that require local CNS-directed therapy, or increasing doses of corticosteroids within the prior 2 weeks of first dose of study treatment
* History of severe hypersensitivity reactions to other monoclonal antibodies and/or their excipients
* Known presence of neutralizing anti-atezolizumab antibodies (for patients previously treated with atezolizumab)
* Having out of range laboratory values: creatinine, bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), absolute neutrophil count (ANC), platelet count, hemoglobin
* Impaired cardiac function or clinically significant cardiac disease, including any of the following:

  1. Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (New York Heart Association [NYHA] Grade ≥2), uncontrolled hypertension or clinically significant arrhythmia
  2. QTcF >470 msec on screening (electrocardiogram) ECG using Fridericia's formula (QTcF) or congenital long QT syndrome
  3. Acute myocardial infarction or unstable angina pectoris
* Known human immunodeficiency virus (HIV), active hepatitis B virus (HBV) or active hepatitis C virus (HCV) infection
* Malignant disease, other than that being treated in this study
* Any medical condition that would, in the Investigator's judgment, prevent participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results
* Active autoimmune disease or a documented history of autoimmune disease
* Participants previously exposed to anti-PD-(L)1 treatment who are not adequately treated for skin rash or had no replacement therapy for endocrinopathies should be excluded
* Participants with a history of drug-induced pneumonitis or current pneumonitis
* Systemic steroid therapy or any immunosuppressive therapy. Topical, inhaled, nasal, and ophthalmic steroids are not prohibited
* Use of live attenuated vaccines against infectious diseases within 4 weeks of the first dose of study treatment. SARS-CoV-2 vaccines authorized for use by the competent local regulatory health authorities for active immunization to prevent COVID 19 are allowed (unless the vaccine is live or live attenuated) and must be given in accordance with the prevailing immunization guidelines.
* Anti-CTLA4, anti-PD-(L)1 treatment within 4 weeks of the first dose of study treatment
* Pre-treatment with anti-CTLA4 antibodies in combination with any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathway
* Presence of Common Terminology Criteria for Adverse Events version 5 (CTCAE v5) ≥Grade 2 toxicity (except alopecia, peripheral neuropathy and ototoxicity, which are excluded if CTCAE v5 ≥Grade 3) due to prior cancer therapy
* Radiotherapy within 2 weeks of the first dose of study treatment, except for palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass. To allow evaluation for response to treatment, participants enrolled in the Phase 2 part must have remaining measurable disease that has not been irradiated
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (22):
- United States (6):
  - Kymab investigational site 1109, Duarte, California
  - Kymab investigational site 1102, New Haven, Connecticut
  - Kymab investigational site 1108, Orlando, Florida
  - Kymab investigational site 1104, Sarasota, Florida
  - Kymab investigational site 1103, Nashville, Tennessee
  - Kymab investigator site 1101, Houston, Texas
- Hungary (2):
  - Kymab investigational site 3601, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Kymab investigational site 3602, Budapest
- Italy (7):
  - Kymab investigational site 3904, Meldola, Forlì-Cesena
  - Kymab investigational site 3906, Candiolo, Torino
  - Kymab investigational site 3901, Milan
  - Kymab investigational site 3903, Milan
  - Kymab investigational site 3902, Napoli
  - Kymab investigational site 3910, Roma
  - Kymab investigational site 3908, Turin
- Kymab investigational site 4801, Siedlce, Masovian Voivodeship, Poland
- Taiwan (2):
  - Kymab investigational site 8806, Changhua, Changhwa
  - Kymab investigational site 8801, Taipei
- United Kingdom (4):
  - Kymab investigational site 4405, London
  - Kymab investigational site 4402, Manchester
  - Kymab investigational site 4404, Oxford
  - Kymab investigational site 4401, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 22 centers in 6 countries. A total of 222 participants, of which 0 were screen failures. Participants were enrolled from 28 January 2019 to 04 August 2023.
Groups:
- Alomfilimab 0.8 mg: Participants received alomfilimab 0.8 mg as a single agent via intravenous (IV) infusion every 3 weeks (Q3W). The participants continued treatment with alomfilimab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed disease progression (PD) per immune-related (i) Response Evaluation Criteria in Solid Tumors (RECIST).
- Alomfilimab 2.4 mg: Participants received alomfilimab 2.4 mg as a single agent via IV infusion Q3W. The participants continued treatment with alomfilimab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 8 mg: Participants received alomfilimab 8 mg as a single agent via IV infusion Q3W. The participants continued treatment with alomfilimab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 24 mg: Participants received alomfilimab 24 mg as a single agent via IV infusion Q3W. The participants continued treatment with alomfilimab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 80 mg: Participants received alomfilimab 80 mg as a single agent via IV infusion Q3W. The participants continued treatment with alomfilimab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 240 mg: Participants received alomfilimab 240 mg as a single agent via IV infusion Q3W. The participants continued treatment with alomfilimab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 0.8 mg + Atezolizumab: Participants received alomfilimab 0.8 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 2.4 mg + Atezolizumab: Participants received alomfilimab 2.4 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 8 mg + Atezolizumab: Participants received alomfilimab 8 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 24 mg + Atezolizumab: Participants received alomfilimab 24 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 80 mg + Atezolizumab: Participants received alomfilimab 80 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer: Anti-PD-(L)1 naïve participants with pancreatic cancer received alomfilimab 2.4 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer: Anti-PD-(L)1 naïve participants with pancreatic cancer received alomfilimab 8 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative Breast Cancer (BC): Anti-PD-(L)1 naïve participants with triple negative BC received alomfilimab 2.4 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC: Anti-PD-(L)1 naïve participants with triple negative BC received alomfilimab 8 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Head and Neck Squamous Cell Carcinoma (HNSCC): Anti-PD-(L)1 naïve participants with HNSCC received alomfilimab 8 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC: Anti-PD-(L)1 naïve participants with HNSCC received alomfilimab 24 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer: Participants with pre-treated pancreatic cancer received alomfilimab 2.4 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer: Participants with pre-treated pancreatic cancer received alomfilimab 8 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC: Participants with pre-treated triple negative BC received alomfilimab 2.4 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC: Participants with pre-treated triple negative BC received alomfilimab 8 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC: Participants with pre-treated HNSCC received alomfilimab 8 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC: Participants with pre-treated HNSCC received alomfilimab 24 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
Period: Overall Study
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative Breast Cancer (BC) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Head and Neck Squamous Cell Carcinoma (HNSCC) | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Started | 4 | 5 | 9 | 8 | 7 | 5 | 5 | 43 | 36 | 9 | 9 | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 9
Treated | 4 | 5 | 9 | 8 | 7 | 5 | 5 | 43 | 36 | 9 | 9 | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
Safety Analysis Set | 4 | 5 | 10 (One participant was planned to receive alomfilimab 8 mg + atezolizumab; however, the actual dose received was alomfilimab 8 mg. For the Safety Analysis Set, this participant was counted under actual dose received (alomfilimab 8 mg).) | 8 | 7 | 5 | 5 | 43 | 35 (One participant was planned to receive alomfilimab 8 mg + atezolizumab; however, the actual dose received was alomfilimab 8 mg. For the Safety Analysis Set, this participant was counted under actual dose received (alomfilimab 8 mg).) | 9 | 9 | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 4 | 4 | 9 | 8 | 7 | 5 | 5 | 40 | 35 | 9 | 9 | 15 | 14 | 6 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 2 | 9
Not completed — Withdrawal of Consent | 2 | 0 | 3 | 0 | 1 | 1 | 0 | 10 | 10 | 3 | 4 | 4 | 4 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 1
Not completed — PD | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study Terminated by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Lost to Follow Up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Death | 2 | 4 | 5 | 6 | 5 | 4 | 5 | 24 | 22 | 6 | 3 | 10 | 10 | 5 | 7 | 2 | 2 | 1 | 1 | 1 | 1 | 2 | 3
Not completed — Miscellaneous | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all participants who were allocated to study drug, regardless of treatment ultimately received.
Groups:
- Alomfilimab 0.8 mg: Participants received alomfilimab 0.8 mg as a single agent via IV infusion Q3W. The participants continued treatment with alomfilimab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC: Anti-PD-(L)1 naïve participants with triple negative BC received alomfilimab 2.4 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC: Anti-PD-(L)1 naïve participants with HNSCC received alomfilimab 8 mg in combination with atezolizumab 1200 mg via IV infusion Q3W. The participants continued treatment with alomfilimab in combination with atezolizumab within this clinical study, as long as they continued to derive benefit from treatment, until the participant experienced unacceptable toxicity or confirmed PD per iRECIST.
- Total: Total of all reporting groups
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Total
Number analyzed (Participants) | 4 | 5 | 9 | 8 | 7 | 5 | 5 | 43 | 36 | 9 | 9 | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 9 | 222
Age, Customized [Count of Participants; unit: Participants]
  >= 18 - 64 years | 2 | 2 | 6 | 2 | 4 | 3 | 2 | 27 | 27 | 5 | 5 | 8 | 5 | 6 | 10 | 3 | 4 | 1 | 0 | 1 | 4 | 3 | 3 | 133
  >= 65 to 84 years | 2 | 3 | 3 | 6 | 3 | 1 | 3 | 16 | 9 | 4 | 4 | 7 | 9 | 1 | 4 | 2 | 1 | 1 | 1 | 0 | 2 | 0 | 6 | 88
  >= 85 years | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 6 | 3 | 3 | 3 | 20 | 20 | 5 | 4 | 6 | 6 | 7 | 14 | 0 | 1 | 0 | 0 | 1 | 6 | 1 | 4 | 118
  Male | 1 | 2 | 7 | 2 | 4 | 2 | 2 | 23 | 16 | 4 | 5 | 9 | 8 | 0 | 0 | 5 | 4 | 2 | 1 | 0 | 0 | 2 | 5 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 9 | 6 | 2 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 28
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 8
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 5 | 8 | 8 | 5 | 5 | 5 | 30 | 28 | 6 | 6 | 14 | 14 | 7 | 13 | 4 | 3 | 2 | 1 | 1 | 3 | 1 | 8 | 181
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Ethnicity was not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a pharmaceutical product, which did not necessarily have a causal relationship with this treatment. An serious AE (SAE) was any AE that:
  * resulted in death;
  * was life-threatening;
  * resulted in inpatient hospitalization or prolongation of existing hospitalization;
  * resulted in a persistent or significant disability/incapacity;
  * resulted in congenital anomaly/birth defect in the offspring of a participant who received IMPs;
  * constituted an important medical event.
  Clinically significant changes in laboratory parameters, vital signs and electrocardiogram results were reported as AEs. A TEAE was defined as an AE observed after starting administration of the specific treatment.
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment; maximum duration of treatment exposure was up to approximately 212 weeks
Population: Safety Analysis Set: all participants who took at least one dose of study drug within the relevant phase. Participants were grouped according to the study drug received at Cycle 1 Day 1 (21-day cycle length).
Measure: Count of Participants; unit: Participants
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 10 | 8 | 7 | 5 | 5 | 43 | 35 | 9 | 9
Participants
  Any TEAEs | 4 | 4 | 8 | 7 | 7 | 5 | 4 | 43 | 34 | 9 | 9
  Any Serious TEAEs | 1 | 1 | 3 | 2 | 3 | 2 | 2 | 17 | 11 | 4 | 3

2. Primary Outcome: Phase 1: Number of Participants Experiencing Dose Changes
Description: Dose changes were defined as infusion interruption and dose reduction.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 10 | 8 | 7 | 5 | 5 | 43 | 35 | 9 | 9
Participants
  Infusion Interruption | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 2
  Dose Reduction | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 1: Absolute Dose Intensity
Description: Absolute dose intensity was calculated as cumulative dose received (mg) / study treatment duration (weeks).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 10 | 8 | 7 | 5 | 5 | 43 | 35 | 9 | 9
mg/week | 0.260 (0.0000) | 0.778 (0.0179) | 2.616 (0.0427) | 7.799 (0.2694) | 26.174 (0.1952) | 76.650 (4.8260) | 0.236 (0.0288) | 0.780 (0.0176) | 2.573 (0.1159) | 7.418 (1.1455) | 25.774 (0.9037)

4. Primary Outcome: Phase 1: Relative Dose Intensity
Description: Relative dose intensity was calculated as the cumulative dose received (mg) / initial planned cumulative dose (mg). Initial planned cumulative dose was calculated as the starting dose multiplied by the scheduled number of administrations within the study treatment duration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 10 | 8 | 7 | 5 | 5 | 43 | 35 | 9 | 9
ratio | 0.988 (0.0189) | 0.978 (0.0179) | 0.979 (0.0179) | 1.015 (0.0835) | 0.980 (0.0058) | 0.958 (0.0610) | 0.884 (0.1071) | 0.978 (0.0202) | 0.963 (0.0432) | 0.928 (0.1422) | 0.967 (0.0316)

5. Primary Outcome: Phase 1: Number of Participants Experiencing Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as a clinically relevant AE or abnormal laboratory value of Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE v5.0) ≥ Grade 3 assessed as unrelated to disease, PD, inter-current illness or concomitant medications, which occurs within the first cycle (21 days) of treatment with alomfilimab as single agent or in combination with atezolizumab during the dose escalation part of the study.
Time Frame: From first dose of study treatment (Day 1) up to 21 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 10 | 8 | 7 | 5 | 5 | 43 | 35 | 9 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Phase 2: Overall Response Rate (ORR) Per RECIST 1.1
Description: ORR was the percentage of participants with a measurable disease at baseline and with a confirmed response of complete response (CR) or partial response (PR) according to RECIST v1.1 as the best response. The response is confirmed by a later scan conducted at least 4 weeks after the initial response is observed. The 95% confidence interval (CI) was calculated using the exact binomial method (Clopper-Pearson).
  CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: From first dose of study treatment (Day 1) up to the end of the long term follow-up, approximately 162 weeks
Population: Full Analysis Set: all participants who were allocated to study drug, regardless of treatment ultimately received. The number of participants analyzed is inclusive of those with measurable disease at baseline only for the purpose of evaluating ORR.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
percentage of participants | 0 [0.0 to 21.8] | 0 [0.0 to 28.5] | 0 [0.0 to 45.9] | 7.1 [0.2 to 36.0] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 52.2] | 33.3 [0.8 to 90.6] | 0 [0.0 to 41.0]

7. Secondary Outcome: Best Overall Response (BOR) Per RECIST 1.1
Description: BOR for each participant was defined as the best confirmed response per RECIST 1.1 among all responses recorded from start of treatment until PD, initiation of new anti-cancer therapy, death, or analysis cut-off date, whichever comes first, with responses of:
  CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
  Stable disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  PD: at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5mm. Unequivocal progression of existing non-target lesions.
  Not evaluable (NE).
Time Frame: From first dose of study treatment (Day 1) up to the end of the long term follow-up, approximately 236 and 162 weeks for Phase 1 and 2, respectively
Population: Full Analysis Set: all participants who were allocated to study drug, regardless of treatment ultimately received.
Measure: Count of Participants; unit: Participants
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 4 | 5 | 9 | 8 | 7 | 5 | 5 | 43 | 36 | 9 | 9 | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 9
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  SD | 1 | 0 | 2 | 2 | 2 | 1 | 3 | 12 | 8 | 1 | 4 | 6 | 0 | 1 | 4 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 3
  PD | 3 | 3 | 7 | 3 | 4 | 4 | 1 | 20 | 22 | 7 | 2 | 9 | 11 | 5 | 8 | 2 | 2 | 1 | 0 | 1 | 3 | 2 | 4
  NE | 0 | 2 | 0 | 3 | 1 | 0 | 1 | 7 | 4 | 0 | 3 | 0 | 3 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 2

8. Secondary Outcome: Progression-free Survival (PFS) Per RECIST 1.1
Description: PFS was calculated as (first documented PD or death due to any cause - first dose date of study drug +1)/30.4375. Participants who were not observed to have progressed or died were censored at the date of the last tumor assessment. Participants who missed two or more sequential assessments were censored at the date of the last tumor assessment before the missed assessments. Participants who started new anti-cancer therapy prior to documented PD were censored at the date of the last tumor assessment prior to the start of the new therapy. Participants who did not have any tumor assessments were censored with a duration of 1 day. PFS was obtained via Kaplan Meier estimation using the Brookmeyer-Crowley method.
  PD: at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5mm. Unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 7
Population: Full Analysis Set: all participants who were allocated to study drug, regardless of treatment ultimately received. The number of participants analyzed is inclusive of those with observed events or participants that were censored for the purpose of evaluating PFS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 4 | 5 | 9 | 8 | 7 | 5 | 5 | 43 | 36 | 9 | 9 | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
months | 2 [2 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 2 [1 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 2 [1 to 6] | 3 [1 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 2 [1 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 1 [1 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 3 [2 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 2 [2 to 4] | 2 [2 to 2] | 2 [1 to 4] | 4 [2 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 2 [1 to 4] | 2 [2 to 2] | 2 [1 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 2 [1 to 4] | 4 [2 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 2 [1 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 2 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 3 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 2 [NA to NA] — Confidence intervals were not calculable due to insufficient event data occurring near the median. | 4 [2 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 2 [2 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 3 [2 to 4]

9. Secondary Outcome: Duration of Response Per RECIST 1.1
Description: Duration of response was calculated as (date of the first documentation of PD or to death due to any cause in the absence of PD - date of the first documentation of unconfirmed objective response [CR or PR] + 1]/30.4375. Participants who were not observed to have progressed or died were censored at the date of the last tumor assessment. Participants who missed two or more sequential assessments were censored at the date of the last tumor assessment before the missed assessments. Participants who started new anti-cancer therapy prior to documented PD were censored at the date of the last tumor assessment prior to the start of the new therapy. Participants with no disease assessment (or only had assessments with response = NE) after first study treatment or have baseline or post-baseline assessments where the RECIST criteria could not be applied had their duration of response time censored. Duration of response was obtained via Kaplan Meier estimation.
Time Frame: as for outcome 7
Population: Full Analysis Set: all participants who were allocated to study drug, regardless of treatment ultimately received. The number of participants analyzed is inclusive of those with observed events or participants that were censored for the purpose of evaluating duration of response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
months |  |  |  |  |  |  | 11 [NA to NA] — Confidence intervals could not be calculated as a single participant was analyzed. | 6 [2.1 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | NA [13.9 to NA] — Median and upper confidence intervals were not calculable due to fewer than 50% events. | 11 [NA to NA] — Confidence intervals could not be calculated as a single participant was analyzed. |  | 2 [NA to NA] — Confidence intervals could not be calculated as a single participant was analyzed. |  |  | 13 [NA to NA] — Confidence intervals could not be calculated as a single participant was analyzed. |  |  |  |  |  |  | NA [NA to NA] — Median and confidence intervals could not be calculated as a single participant was censored. |

10. Secondary Outcome: ORR Per iRECIST
Description: RECIST 1.1 has been modified to take into consideration the unique response kinetics which have been observed with immunotherapy in some patients where responses to immune therapies may occur after progression has been assessed. ORR was the percentage of participants with a measurable disease at baseline and with a confirmed response of complete immune-response (iCR) or partial immune-response (iPR) according to iRECIST as the best response. The 95% CI was calculated using the exact binomial method (Clopper-Pearson).
  iCR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  iPR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: as for outcome 7
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 4 | 5 | 8 | 8 | 7 | 5 | 4 | 41 | 36 | 9 | 9 | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
percentage of participants | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 33.6] | 0 [0.0 to 52.2] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2] | 9.3 [3.1 to 26.1] | 5.6 [0.8 to 21.4] | 11.1 [0.3 to 48.2] | 0 [0.0 to 45.9] | 0 [0.0 to 23.2] | 0 [0.0 to 30.8] | 0 [0.0 to 45.9] | 7.1 [0.2 to 38.5] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 97.5] | 0 [0.0 to 52.2] | 33.3 [2.5 to 100.0] | 0 [0.0 to 41.0]

11. Secondary Outcome: PFS Per iRECIST
Description: PFS was calculated as (first documented iPD or death due to any cause - first dose date of study drug +1)/30.4375. Participants who were not observed to have progressed or died were censored at the date of the last tumor assessment. Participants who missed two or more sequential assessments were censored at the date of the last tumor assessment before the missed assessments. Participants who started new anti-cancer therapy prior to documented PD were censored at the date of the last tumor assessment prior to the start of the new therapy. Participants who did not have any tumor assessments were censored with a duration of 1 day. PFS was obtained via Kaplan Meier estimation using the Brookmeyer-Crowley method.
  iPD: at least a 20% increase in the sum of diameters of target lesions. The sum must also demonstrate an increase of at least 5mm. Unequivocal progression of existing non-target lesions.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 4 | 5 | 9 | 8 | 7 | 5 | 5 | 43 | 36 | 9 | 9 | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
months | 7 [NA to NA] — Confidence intervals could not be calculated as a single participant had observed events. | 10 [4.2 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 10 [3.4 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 6 [3.3 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 6 [2.7 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 6 [3.4 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 4 [2.5 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 7 [5.5 to 10.0] | 5 [2.8 to 9.9] | 3 [1.8 to 4.0] | 5 [4.6 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 5 [2.5 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 5 [2.7 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 4 [2.6 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 10 [1.7 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 5 [5.0 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | 4 [1.5 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median. | NA [NA to NA] — Median and confidence intervals could not be calculated as two participants were censored. | 10 [NA to NA] — Confidence intervals could not be calculated as a single participant had observed events. | 17 [NA to NA] — Confidence intervals could not be calculated as a single participant had observed events. | 12 [NA to NA] — Confidence intervals could not be calculated as a single participant had observed events. | NA [NA to NA] — Median and confidence intervals could not be calculated as three participants were censored. | 6 [2.6 to NA] — Upper confidence interval was not calculable due to insufficient event data occurring above the median.

12. Secondary Outcome: Phase 1: ORR Per RECIST 1.1
Description: ORR was the percentage of participants with a measurable disease at baseline and with a confirmed response of CR or PR according to RECIST v1.1 as the best response. The response is confirmed by a later scan conducted at least 4 weeks after the initial response is observed. The 95% CI was calculated using the exact binomial method (Clopper-Pearson).
  CR: disappearance of all target and non-target lesions. Any pathological lymph nodes (whether target or non-target) must have had a reduction in short axis to < 10 mm. All lymph nodes must have been non-pathological in size (< 10mm short axis).
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the Baseline sum diameters.
Time Frame: From first dose of study treatment (Day 1) up to the end of the long term follow-up, approximately 236 weeks
Population: Full Analysis Set: all participants who were allocated to study drug, regardless of treatment ultimately received. Inclusive of participants with measurable disease at baseline only.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 8 | 8 | 7 | 5 | 4 | 41 | 36 | 9 | 9
percentage of participants | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 33.6] | 0 [0.0 to 52.2] | 0 [0.0 to 45.9] | 0 [0.0 to 52.2] | 0 [0.0 to 60.2] | 9.3 [3.1 to 26.1] | 5.6 [0.8 to 20.8] | 11.1 [0.3 to 48.2] | 0 [0.0 to 45.9]

13. Secondary Outcome: Overall Survival Rate at 12 and 24 Months
Description: Overall Survival rate was defined as the proportion of participants that had known survival status. Overall survival rate was obtained via Kaplan Meier estimation using the complimentary log-log transformation method.
Time Frame: Months 12 and 24
Population: Full Analysis Set: all participants who were allocated to study drug, regardless of treatment ultimately received.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 4 | 5 | 9 | 8 | 7 | 5 | 5 | 43 | 36 | 9 | 9 | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 9
proportion of participants
  12 months | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 12 months. | 0.2 [0.01 to 0.58] | 0.4 [0.10 to 0.73] | 0.3 [0.04 to 0.56] | 0.4 [0.10 to 0.73] | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 12 months. | 0.4 [0.05 to 0.75] | 0.4 [0.27 to 0.60] | 0.4 [0.22 to 0.57] | 0.2 [0.01 to 0.64] | 0.5 [0.12 to 0.82] | 0.2 [0.03 to 0.47] | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 12 months. | 0.6 [0.17 to 0.84] | 0.7 [0.38 to 0.88] | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 12 months. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | 0.3 [0.01 to 0.77] | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint.
  24 months | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 24 months. | 0.2 [0.01 to 0.58] | 0.3 [0.04 to 0.61] | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 24 months. | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 24 months. | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 24 months. | 0.3 [0.13 to 0.43] | 0.3 [0.11 to 0.44] | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 24 months. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 24 months. | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 24 months. | 0.2 [0.01 to 0.56] | 0.4 [0.13 to 0.66] | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 24 months. | 0.0 [NA to NA] — Confidence intervals could not be calculated as no participants had known survival status at 24 months. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint. | NA [NA to NA] — Number and confidence intervals could not be calculated as all participants were not alive or survival status was unknown at this timepoint.

14. Secondary Outcome: Phase 2: Number of Participants Experiencing TEAEs
Description: An AE was any untoward medical occurrence in a participant administered a pharmaceutical product, which did not necessarily have a causal relationship with this treatment. An SAE was any AE that:
  * resulted in death;
  * was life-threatening;
  * resulted in inpatient hospitalization or prolongation of existing hospitalization;
  * resulted in a persistent or significant disability/incapacity;
  * resulted in congenital anomaly/birth defect in the offspring of a participant who received IMPs;
  * constituted an important medical event.
  Clinically significant changes in laboratory parameters, vital signs and electrocardiogram results were reported as AEs. A TEAE was defined as an AE observed after starting administration of the specific treatment.
Time Frame: From first dose of study treatment (Day 1) up to 30 days post last dose of study treatment; maximum duration of treatment exposure was up to approximately 86 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
Participants
  Any TEAEs | 15 | 13 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
  Any Serious TEAEs | 6 | 2 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 4

15. Secondary Outcome: Phase 2: Number of Participants Experiencing Dose Changes
Description: Dose changes were defined as infusion interruption and dose reduction.
Time Frame: as for outcome 14
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
Participants
  Infusion Interruption | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Dose Reduction | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Phase 2: Absolute Dose Intensity
Description: Absolute dose intensity was calculated as cumulative dose received (mg) / study treatment duration (weeks).
Time Frame: as for outcome 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/week
Arm/Group | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
mg/week | 0.778 (0.0540) | 2.559 (0.1712) | 0.777 (0.0111) | 2.536 (0.1628) | 2.366 (0.3577) | 6.818 (2.3926) | 0.775 (0.0212) | 2.640 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 0.760 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 2.607 (0.0841) | 2.613 (0.0551) | 7.794 (0.1676)

17. Secondary Outcome: Phase 2: Relative Dose Intensity
Description: as for outcome 4
Time Frame: as for outcome 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 15 | 14 | 7 | 14 | 5 | 5 | 2 | 1 | 1 | 6 | 3 | 8
ratio | 0.973 (0.0660) | 0.956 (0.0638) | 0.976 (0.0113) | 1.014 (0.1256) | 0.886 (0.1316) | 0.980 (0.0274) | 0.975 (0.0212) | 0.990 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 0.960 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 0.977 (0.0333) | 0.980 (0.0200) | 0.973 (0.0191)

18. Secondary Outcome: Phase 1: Maximum Concentration (Cmax) of Alomfilimab
Description: The serum pharmacokinetics (PK) of alomfilimab were characterized using non-compartmental analysis (NCA). Nominal times of sample collections were used for the NCA. All below limit of quantification (BLQ) values were set to 0 units.
Time Frame: Cycles 1 and 3 Day 1 pre-infusion to 336 hours post-infusion start (21 day cycle length)
Population: PK Evaluable Set: consisted of all participants who had sufficient concentration-time data within the relevant phase to permit calculation of PK parameters for alomfilimab.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 7 | 5 | 5 | 35 | 29 | 8 | 9
ug/mL
  Cycle 1 | 0.3022 (0.12476) | 0.9773 (0.29919) | 3.3327 (0.95752) | 8.7301 (2.84671) | 33.7844 (12.98646) | 124.4294 (79.79754) | 0.3339 (0.17905) | 1.1201 (0.66885) | 3.3476 (1.23416) | 8.2597 (2.75396) | 31.4793 (10.38008)
  Cycle 3: number analyzed (Participants) | 3 | 2 | 7 | 3 | 5 | 2 | 3 | 25 | 21 | 5 | 6
  Cycle 3 | 0.2671 (0.06805) | 1.2029 (0.24583) | 3.7461 (0.86853) | 30.5647 (39.72256) | 43.8045 (14.07259) | 141.8131 (62.54794) | 0.2840 (0.24914) | 1.6449 (3.01380) | 9.5099 (28.23379) | 10.2883 (3.86029) | 51.6622 (41.65071)

19. Secondary Outcome: Phase 1: Half-life (t1/2) of Alomfilimab
Description: The serum PK of alomfilimab were characterized using NCA. Nominal times of sample collections were used for the NCA. All BLQ values were set to 0 units.
Time Frame: Cycles 1 and 3 Day 1 pre-infusion to 336 hours post-infusion start (21 day cycle length)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab
Number analyzed (Participants) | 4 | 5 | 9 | 8 | 7 | 5 | 4 | 36 | 30 | 8 | 9
hours
  Cycle 1 | 42.7633 (20.84762) | 72.2276 (9.56084) | 149.0872 (55.14152) | 226.2922 (75.20291) | 377.5444 (126.28273) | 356.4297 (109.96450) | 37.4777 (3.96733) | 93.0339 (33.82676) | 165.8783 (89.07566) | 174.9685 (79.39134) | 300.0089 (113.49910)
  Cycle 3: number analyzed (Participants) | 0 | 1 | 5 | 2 | 5 | 1 | 0 | 15 | 14 | 2 | 5
  Cycle 3 |  | 80.3268 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 215.6472 (98.90118) | 358.6064 (143.16181) | 342.6067 (193.81667) | 273.6673 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |  | 116.0599 (42.16269) | 202.0099 (78.48781) | 230.5514 (103.13822) | 440.0235 (236.99886)

20. Secondary Outcome: Number of Participants Experiencing Anti-drug Antibodies (ADA) at Anytime
Description: Detection of ADA was assessed from blood samples taken during the study using validated bioanalytical methods. The number of participants who developed detectable anti-alomfilimab or anti-atezolizumab antibodies during any cycle or the safety follow-up period (SFUP) was calculated.
Time Frame: Phase 1: pre-infusion at all cycles (up to 69 cycles) + 90 days SFUP; Phase 2: pre-infusion at all cycles (up to 28 cycles) + 90 day SFUP (21 day cycle length)
Population: Anti-drug Antibody Evaluable Set: consisted of all participants who received at least one dose of alomfilimab or atezolizumab and had ADA results available for analysis within the relevant phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 4 | 3 | 8 | 8 | 7 | 5 | 5 | 36 | 34 | 8 | 6 | 13 | 11 | 6 | 12 | 5 | 3 | 1 | 1 | 0 | 6 | 3 | 7
Participants
  ≥ 1 Positive Anti-alomfilimab Antibodies Result: number analyzed (Participants) | 4 | 3 | 8 | 8 | 7 | 5 | 5 | 36 | 34 | 8 | 6 | 13 | 11 | 6 | 12 | 4 | 0 | 1 | 1 | 0 | 6 | 3 | 0
  ≥ 1 Positive Anti-alomfilimab Antibodies Result | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 9 | 8 | 0 | 0 | 1 | 2 | 1 | 0 | 3 |  | 1 | 0 |  | 0 | 1 |
  ≥ 1 Positive Anti-atezolizumab Antibodies Result: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 36 | 34 | 8 | 6 | 13 | 11 | 6 | 12 | 5 | 3 | 1 | 1 | 0 | 6 | 3 | 7
  ≥ 1 Positive Anti-atezolizumab Antibodies Result |  |  |  |  |  |  | 1 | 8 | 8 | 4 | 1 | 5 | 2 | 1 | 0 | 1 | 0 | 0 | 0 |  | 0 | 1 | 1

21. Secondary Outcome: Change From Baseline in Tumor-infiltrating Lymphocytes Per mm^2 at Cycle 2 Day 8
Description: Biological samples (e.g., archived and fresh tumor samples or blood samples) were collected for analysis of responsive biomarkers.
  The summary of change in the following markers were calculated:
  * FOXP3-ICOS double-positive cells per mm^2 in the Tumor
  * CD8-positive cells per mm^2 in the tumor
  * CD8-positive cells per mm^2 in the invasive margin.
Time Frame: Baseline and Cycle 2 Day 8 (21 day cycle length)
Population: Biomarker Evaluable Set: consisted of all participants who received at least one dose of study drug and had at least one of ICOS, FOXP3 and CD8 cells results available for analysis within the relevant phase.
Measure: Mean (Standard Deviation); unit: cells per mm^2
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
Number analyzed (Participants) | 2 | 3 | 7 | 3 | 5 | 3 | 3 | 16 | 16 | 3 | 3 | 8 | 5 | 4 | 8 | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 3
cells per mm^2
  FOXP3-ICOS double-positive cells per mm^2 in the tumor: number analyzed (Participants) | 2 | 2 | 6 | 3 | 5 | 3 | 3 | 16 | 14 | 3 | 3 | 6 | 5 | 4 | 8 | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 3
  FOXP3-ICOS double-positive cells per mm^2 in the tumor | 0.275 (5.5649) | 21.905 (30.1015) | -50.323 (42.9514) | -42.210 (26.6714) | -29.318 (28.0896) | -67.160 (59.7524) | -18.860 (33.2369) | -129.334 (118.3340) | -90.589 (115.9495) | -117.610 (174.4591) | -3.653 (6.5269) | -58.865 (65.7823) | -45.618 (34.5880) | -51.293 (56.8048) | -76.331 (63.0946) | -437.660 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | -518.975 (668.5624) |  | -31.120 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |  | -149.445 (137.0019) | -197.940 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | -397.437 (307.3676)
  CD8-positive cells per mm^2 in the tumor: number analyzed (Participants) | 1 | 3 | 7 | 3 | 5 | 3 | 3 | 14 | 16 | 3 | 2 | 8 | 5 | 3 | 8 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 3
  CD8-positive cells per mm^2 in the tumor | -449.920 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 448.833 (443.5399) | 47.126 (294.7947) | -105.110 (190.2826) | -11.532 (169.8503) | -371.857 (884.7449) | -218.017 (282.9603) | 111.154 (939.3540) | 174.339 (693.8745) | 300.433 (325.6656) | 21.925 (56.3211) | 202.501 (588.9525) | -63.528 (65.5904) | 318.470 (385.7782) | 320.923 (685.1093) | -116.950 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | -1009.800 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |  | -34.840 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |  | 181.120 (147.3752) | -39.600 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 171.170 (293.3937)
  CD8-positive cells per mm^2 in the invasive margin: number analyzed (Participants) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CD8-positive cells per mm^2 in the invasive margin |  |  | -229.600 (114.8200) |  | 336.140 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |  | -422.680 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |  |  | -163.910 (NA) — Standard deviation could not be calculated as a single participant was analyzed. |  |  |  |  |  |  |  |  |  |  |  |  |

ADVERSE EVENTS:
Time Frame: AEs: up to 30 days post last dose of study treatment, a maximum of approximately 216 and 90 weeks for Phase 1 and 2, respectively; All-cause mortality: up to the end of the long term follow-up, a maximum of approximately 236 and 162 weeks for Phase 1 and 2, respectively
Description: AEs are presented per the Safety Analysis Set with participants grouped according to the study drug received at Cycle 1 Day 1 (21-day cycle length). All-cause mortality is presented per the Full Analysis Set.
Arm/Group | Alomfilimab 0.8 mg | Alomfilimab 2.4 mg | Alomfilimab 8 mg | Alomfilimab 24 mg | Alomfilimab 80 mg | Alomfilimab 240 mg | Alomfilimab 0.8 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab | Alomfilimab 8 mg + Atezolizumab | Alomfilimab 24 mg + Atezolizumab | Alomfilimab 80 mg + Atezolizumab | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC
All-Cause Mortality (participants affected / at risk) | 2/4 | 4/5 | 5/9 | 7/8 | 5/7 | 4/5 | 5/5 | 24/43 | 22/36 | 6/9 | 3/9 | 10/15 | 10/14 | 5/7 | 7/14 | 3/5 | 2/5 | 1/2 | 1/1 | 1/1 | 1/6 | 2/3 | 4/9
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/5 | 3/10 | 2/8 | 3/7 | 2/5 | 2/5 | 17/43 | 11/35 | 4/9 | 3/9 | 6/15 | 2/14 | 1/7 | 2/14 | 1/5 | 1/5 | 1/2 | 0/1 | 0/1 | 2/6 | 1/3 | 4/8
Other Adverse Events (participants affected / at risk) | 4/4 | 4/5 | 7/10 | 7/8 | 7/7 | 5/5 | 4/5 | 39/43 | 34/35 | 9/9 | 9/9 | 15/15 | 13/14 | 7/7 | 14/14 | 5/5 | 5/5 | 2/2 | 1/1 | 1/1 | 6/6 | 2/3 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alomfilimab 0.8 mg (N=4) | Alomfilimab 2.4 mg (N=5) | Alomfilimab 8 mg (N=10) | Alomfilimab 24 mg (N=8) | Alomfilimab 80 mg (N=7) | Alomfilimab 240 mg (N=5) | Alomfilimab 0.8 mg + Atezolizumab (N=5) | Alomfilimab 2.4 mg + Atezolizumab (N=43) | Alomfilimab 8 mg + Atezolizumab (N=35) | Alomfilimab 24 mg + Atezolizumab (N=9) | Alomfilimab 80 mg + Atezolizumab (N=9) | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer (N=15) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer (N=14) | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC (N=7) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC (N=14) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC (N=5) | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC (N=5) | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer (N=2) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer (N=1) | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC (N=1) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC (N=6) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC (N=3) | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alomfilimab 0.8 mg (N=4) | Alomfilimab 2.4 mg (N=5) | Alomfilimab 8 mg (N=10) | Alomfilimab 24 mg (N=8) | Alomfilimab 80 mg (N=7) | Alomfilimab 240 mg (N=5) | Alomfilimab 0.8 mg + Atezolizumab (N=5) | Alomfilimab 2.4 mg + Atezolizumab (N=43) | Alomfilimab 8 mg + Atezolizumab (N=35) | Alomfilimab 24 mg + Atezolizumab (N=9) | Alomfilimab 80 mg + Atezolizumab (N=9) | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer (N=15) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Pancreatic Cancer (N=14) | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC (N=7) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve Triple Negative BC (N=14) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC (N=5) | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Naïve HNSCC (N=5) | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer (N=2) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Pancreatic Cancer (N=1) | Alomfilimab 2.4 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC (N=1) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated Triple Negative BC (N=6) | Alomfilimab 8 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC (N=3) | Alomfilimab 24 mg + Atezolizumab in Anti-PD-(L)1 Pre-treated HNSCC (N=8)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (4) | 2 (3) | 0 (0) | 9 (15) | 11 (20) | 3 (3) | 3 (5) | 5 (8) | 1 (2) | 0 (0) | 3 (6) | 1 (2) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (3) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 2 (4) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 5 (5) | 2 (4) | 2 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 5 (9) | 5 (7) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (3) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 4 (6) | 3 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 8 (10) | 10 (11) | 1 (1) | 2 (2) | 0 (0) | 6 (7) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 9 (15) | 10 (13) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (7) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 9 (14) | 8 (8) | 5 (5) | 6 (6) | 4 (7) | 2 (3) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 3 (5) | 2 (5) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4) | 5 (6) | 5 (10) | 1 (1) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (6) | 2 (3) | 1 (3) | 0 (0) | 2 (3) | 3 (6) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 7 (9) | 1 (1) | 0 (0) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 4 (6) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (6) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour cavitation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmetria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 3 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Hemianopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemianopia homonymous (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 7 (10) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 8 (11) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 4 (4) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT03829501/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/01/NCT03829501/SAP_001.pdf